CLINICAL TRIAL: NCT01653145
Title: Behavioral Response to Short-term (Two-day) Positive Energy Balance Through Overfeeding (ENERGY I)
Brief Title: Positive Energy I Through Overfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: PBRC 10017
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Appetite; Satiety
MeSH Terms: conditions — Obesity | interventions — Carbohydrates; Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diet A (Active Comparator): Low Fat High Energy Density (1.6 kcal/g)-50% Fat, 35% Carbohydrate, and 15% Protein
  Interventions: Other: Diet A; Other: Diet B; Other: Diet C
- Diet B (Active Comparator): High Fat Low Energy Density (1.05 kcal/g)-50% Fat, 35% Carbohydrate, and 15% Protein
  Interventions: Other: Diet A; Other: Diet B; Other: Diet C
- Diet C (Active Comparator): High Carbohydrate Low Energy Density (1.05 kcal/g)-20% Fat, 65% Carbohydrate, 15% Protein
  Interventions: Other: Diet A; Other: Diet B; Other: Diet C

INTERVENTIONS:
Other: Diet A — Dietary
  Other Names: Low Fat High Energy Density (1.6 kcal/g)-50% Fat, 35% Carbohydrate, and 15% Protein
Other: Diet B — Dietary
  Other Names: High Fat Low Energy Density (1.05 kcal/g)-50% Fat, 35% Carbohydrate, and 15% Protein
Other: Diet C — Dietary
  Other Names: High Carbohydrate Low Energy Density (1.05 kcal/g)-20% Fat, 65% Carbohydrate, 15% Protein

SUMMARY:
The purpose of this trial is to examine the metabolic and behavioral effects of a positive energy balance induced by adding food to the usual level of activity.

It is hypothesized that: 1) food intake will not differ significantly after 2 days of positive energy balance induced by a high carbohydrate vs. high fat diet when both diets are low in energy density, and 2) food intake will be higher after a positive energy balance induced by a high fat/high energy dense diet vs. a high fat/low energy dense diet.

DETAILED DESCRIPTION:
The purpose of this trial is to examine the metabolic and behavioral effects of a positive energy balance induced by adding food to the usual level of activity. During this study, we will induce a positive energy balance for two days by increasing food intake to 140% of baseline energy requirements and keeping energy expenditure constant. The following three diets, which vary in dietary fat and energy density (kcal/g), will be used to induce the positive energy balance in a within subjects or cross over design: 1) high fat/high energy density, 2) high fat/low energy density, and 3) high carbohydrate/low energy density. Food intake and activity will be measured for 4 days after each diet to quantify the response to positive energy balance and manipulation of dietary fat and energy density.

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 18 and 50, inclusive, if you are a male or between the ages of 18 and 45, inclusive, if you are a female.
* Your body mass index (BMI) is between 20 and 40 kg/m², inclusive.
* For females, if you have regular menstrual periods, with no less than 28 day cycles. Monophasic birth control pills, copper IUD, Ortho Evra patch, NuvaRing or complete hysterectomy are also acceptable.

Exclusion Criteria:

* You have a chronic disease that affects body weight, appetite, or metabolism, such as diabetes and cardiovascular disease.
* You have irregular menstrual cycles, had a partial hysterectomy (still maintain ovaries), or use an IUD not made of copper.
* You use prescriptions or over-the-counter medications or herbal products that affect metabolism or body weight (e.g. weight loss medications such as sibutramine, or orlistat).
* You use a birth control pill that isn't monophasic or you receive Depro-Provera injections.
* You have barriers to completing the study, such as work or family commitments.
* You have symptoms of depression or excessive dietary restraint.
* You use tobacco products.
* You exercise more than 1 hour per day, 5 or more days per week.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Energy Intake | 4 days following the 2 day overfeeding
  Food intake will be measured for 4 days after positive energy balance by directly weighing foods before and after ad libitum lunch and dinner. All food intake testes will occur while the participant resides in the inpatient unit.

SECONDARY OUTCOMES:
Energy Expenditure | 4 days following 2 days of overfeeding
  Armbands were worn by participants throughout the protocol to quantify changes in activity levels and energy expenditure to positive energy balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Apolzan JW, Bray GA, Hamilton MT, Zderic TW, Han H, Champagne CM, Shepard D, Martin CK. Short-term overeating results in incomplete energy intake compensation regardless of energy density or macronutrient composition. Obesity (Silver Spring). 2014 Jan;22(1):119-30. doi: 10.1002/oby.20587. Epub 2013 Sep 10. PMID 23913807